CLINICAL TRIAL: NCT07357519
Title: A Phase 1/2, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, -Radiation Dosimetry, and Preliminary Anti-Neoplastic Activity of LNTH-2403, a LRRC15-targeted 177Lutetium-labeled Monoclonal Antibody, in Participants With Relapsed / Refractory Osteosarcoma
Brief Title: Lu-TARGO (177Lu-TARGeted Osteosarcoma Therapy)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNTH2403-1301
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Relapsed / Refractory Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Clinical Trials, Phase II as Topic

STUDY DESIGN:
Intervention Model Description: Phase 1 will evaluate escalating doses of LNTH-2403 administered once every 8 weeks, with the potential to explore other dosing schedules based on observed radiation dosimetry and PK parameters and safety and tolerability data.
  Phase 2 will evaluate LNTH-2403 as a single agent in participants with R/R osteosarcoma at the recommended phase 2 dose (RP2D).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1- Escalating doses of LNTH-2403 administered once every 8 weeks (Experimental): Phase 1 will evaluate escalating doses of LNTH-2403 administered once every 8 weeks, with the potential to explore other dosing schedules based on observed radiation dosimetry and PK parameters and safety and tolerability data.
  Interventions: Drug: LNTH2403 Phase 1 dose
- Phase 2 will evaluate LNTH-2403 as a single agent at the recommended phase 2 dose (Experimental): Phase 2 will evaluate LNTH-2403 as a single agent in participants with R/R osteosarcoma at the recommended phase 2 dose (RP2D).
  Interventions: Drug: Phase 2; LNTH2403 a single agent recommended phase 2 dose (RP2D).

INTERVENTIONS:
Drug: LNTH2403 Phase 1 dose — LNTH-2403 administered once every 8 weeks, with the potential to explore other dosing schedules based on observed radiation dosimetry and PK parameters and safety and tolerability data.
  Arms: Phase 1- Escalating doses of LNTH-2403 administered once every 8 weeks
Drug: Phase 2; LNTH2403 a single agent recommended phase 2 dose (RP2D). — Once the RP2D is selected, phase 2 will commence
  Arms: Phase 2 will evaluate LNTH-2403 as a single agent at the recommended phase 2 dose

SUMMARY:
This is a multi-center, non-randomized, open-label, dosimetry and dose-escalation, cohort-expansion study of LNTH-2403 administered to subjects with relapsed / refractory (R/R) osteosarcoma. This study consists of 2 phases: (1) a dosimetry and dose escalation phase; and (2) a cohort expansion phase.

ELIGIBILITY:
Inclusion Criteria: Participants must meet all the following criteria to be enrolled in the study

1. Histopathologic documented diagnosis of R/R osteosarcoma
2. Must have disease characterized by at least one of the following (Participants meeting only (b.), only (c.), or only (b. and c.) must be discussed with and receive written approval from the Sponsor to qualify).

   1. Measurable as defined in RECIST 1.1
   2. Evaluable non-measurable disease as per RECIST 1.1
   3. Bone only without a soft tissue component: must be 18F-FDG-PET avid and evaluable by serial 18F-FDG-PET imaging studies.
3. Age: a. First Cohort in Phase 1: ≥ 18 years-of-age at the time of signature of the main study ICF. b. Second and subsequent cohorts, in Phase 1 and all participants in Phase 2: ≥12years-of-age at the time of signature of the main ICF.
4. Performance Status:

   1. Eastern Cooperative Oncology Group (ECOG) Performance Score (PS): 0 - 2
   2. Lansky PS ≥ 50.
5. Body weight: ≥ 30 kg.
6. Tumor biopsies; Fresh or Archival
7. Progression following at least one course of chemotherapy, which includes neoadjuvant / perioperative systemic therapy.
8. All adverse events (AEs) related to prior therapies (chemotherapy / systemic therapies, radiation, surgery) must have resolved to Grade 1 or baseline
9. Organ Function
10. Pregnancy Women of Child-Bearing Potential (WOCBP) must have a negative serum pregnancy test result at screening
11. Contraception- Male participants with a WOCBP partner must use 2 forms of acceptable contraception
12. Written informed consent and/or assent must be obtained according to local guidelines and signed and dated by the participant, parent, and/or legal guardian prior to the performance of any study-specific procedures, sampling, or analyses

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from the study

1. Known allergies, hypersensitivity, or intolerance to LNTH-2403 and/or its excipients
2. Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the investigator's opinion, may affect the participant's safety, compliance with the study, or otherwise impair the assessment of study results
3. Concurrent treatment with any other anti-neoplastic agents, including localized radiation therapy
4. Known active infection
5. Participation in an interventional study of another investigational agent
6. Prior therapies or diagnostics
7. Active prior or concurrent malignancy: immunoglobulin),
8. Known active liver disease from any cause, Hepatitis A Virus
9. Known to be human immunodeficiency virus (HIV) positive
10. Clinically relevant cardiovascular disease
11. Receipt of live vaccine within the 30 days prior to the first dose o
12. A female participant who is pregnant or breastfeeding
13. Major surgical procedure within 28 days of the first dose of LNTH-2403.
14. Participant is unwilling or unable to comply with the scheduled visits, drug administration plan, laboratory tests, or other study procedures and study restrictions

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
To identify the maximum tolerated dose (MTD) of LNTH-2403 in participants with R/R osteosarcoma (Ph1) | From enrollment to the end of treatment at 8 weeks
  Incidence of DLTs during the first 8 weeks (DLT evaluation window) after the first dose of LNTH-2403
To evaluate the safety and tolerability profile of LNTH-2403 in participants with R/R osteosarcoma (Ph1) | From enrollment to the end of treatment at 8 weeks
  Type, frequency, severity, timing, and relationship to LNTH-2403 of all Treatment-emergent adverse event, (TEAEs) and Serious adverse events, (SAEs)
To assess the preliminary anti-neoplastic activity of LNTH-2403 in participants with R/R osteosarcoma (Ph2) | From enrollment to Event-Free Survival (EFS) at 4 months
  Event-Free Survival (EFS) at 4 months

SECONDARY OUTCOMES:
To assess the preliminary anti-neoplastic activity of LNTH-2403 in participants with R/R osteosarcoma (Ph1) | 8 weeks
  Event-Free Survival (EFS) at 8 weeks
To describe the safety and tolerability profile of LNTH-2403 in participants with R/R osteosarcoma (Ph2) | 4 months
  Type, frequency, severity, timing, and relationship to LNTH-2403 of any TEAEs and SAEs

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States